CLINICAL TRIAL: NCT02271672
Title: Effect of the XP1000 RF Therapy on Waist Circumference Reduction
Brief Title: XP1000 RF Therapy on Waist Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XP1000RF
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Circumferential Reduction; Waist Circumferential Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XP1000 RF group (Experimental): Subjects in the XP1000 RF group will be treated with the XP1000 RF device.
  Interventions: Device: XP1000 RF
- Sham group (Sham Comparator): Subjects in the Sham group will be treated with the sham XP1000 RF device.
  Interventions: Device: sham XP1000 RF

INTERVENTIONS:
Device: XP1000 RF — Treatment of adipose tissue within the fat layer with XP1000 RF.
  Arms: XP1000 RF group
Device: sham XP1000 RF — Treatment of adipose tissue within the fat layer with XP1000 RF.
  Arms: Sham group

SUMMARY:
This study was designed to demonstrate safety and efficacy of the XP1000 RF for non-invasive temporary reduction of waist circumference by disruption of adipocyte cells.

DETAILED DESCRIPTION:
This study is a prospective, double-blinded, randomized, two-arm sham-controlled study of circumferential waist reduction following 4 treatment sessions delivered once a week over a 4-week period. The objective of the study is to demonstrate the effectiveness of the treatment after 30-day and 90-day Follow Up in achieving waist circumference reduction of ≥3 cm across the waist line relative to the base line assessment and their mean waist circumferential reduction is ≥1 cm than the average circumferential reduction of sham group.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 20 to 35 kg/m2.
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring and/or weight loss during study participation.
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation.

Exclusion Criteria:

* Implanted electronic device such as a cardiac pacemaker, bladder stimulator, spinal cord stimulator or electrodes for a myoelectric prosthesis, etc.
* Diabetics dependent on insulin or oral hypoglycemic medications
* Known cardiovascular disease such as arrhythmias, congestive heart failure
* Cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers.
* Prior surgical interventions for body sculpting of abdomen such as liposuction
* Medical, physical or other contraindications for body sculpting/ weight loss
* Current use of medication known to affect weight levels and/or cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent
* Any medical condition known to affect weight levels and/or to cause bloating or swelling
* Active infection, wound or other external trauma to the area to be treated
* Pregnant, breast feeding, or planning pregnant before the end of the study
* Serious mental health illness
* Active or recurrent cancer or current chemotherapy and/or radiation treatment
* Negative affection to heat

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Waist Circumferential reduction | 30 days follow follow up after 4 once-a-week treatments
  The primary efficacy outcome measure is set to be a minimum of 80% of subjects in the XP1000 RF group at 30-day follow up evaluation to show waist circumference reduction of ≥3 cm across the waist line relative to the base line assessment and their mean waist circumferential reduction is ≥1 cm than the average circumferential reduction of Sham group.

SECONDARY OUTCOMES:
Adverse Events | 1 month follow up
  Absence of adverse events (AE) associated with the treatment procedure. Safety evaluations of skin reaction in the treatment area would be conducted at every treatment and follow up visits
Adverse Events | 3 months follow up
  Absence of adverse events (AE) associated with the treatment procedure. Safety evaluations of skin reaction in the treatment area would be conducted at every treatment and follow up visits

CONTACTS AND LOCATIONS:
Overall Officials: Radina Denkova, MD, Principal Investigator — Aesthe Beauty Clinic